CLINICAL TRIAL: NCT05952414
Title: The Power of Self-efficacy-based Interventions in Fostering Caring Self-efficacy and Overcoming Job-related Stress and Perceived Stigma Among Psychiatric Nurses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mahmoud Khedr, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0019
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Caring Efficacy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Experimental: Intervention group Group one (study group, 40 nurses): received self-efficacy-based interventions.
  Interventions: Behavioral: self-efficacy-based interventions
- Control group (No Intervention): Group two(the control group, 40 nurses):act as a control group/ waiting list

INTERVENTIONS:
Behavioral: self-efficacy-based interventions — The intervention aims at increasing self-efficacy and consists of Cognitive Behavioural Therapy (CBT)-based exercises related to sources of self-efficacy beliefs: 1) mastery experiences, 2) vicarious experiences, 3) verbal persuasions, and 4) emotional and physiological states.
  Arms: Intervention group

SUMMARY:
People with high self-efficacy set goals to challenge and improve their task achievement rate; however, people with low self-efficacy tend to have fluctuation in their ways of thinking, which results in dampened spirits. Self-efficacy affects mental health. Therefore, psychiatric nurses' achievements that affect their self-efficacy may differ from those of general workers or other nurses. In such a situation, psychiatric nurses feel that uncertainty of care and an unmotivated appearance of the patient can lead to reduced self-efficacy. Consequently, nurses are likely to give up active involvement with patients who will not be leaving the hospital.

DETAILED DESCRIPTION:
The intervention aims at increasing self-efficacy and consists of Cognitive Behavioural Therapy (CBT)-based exercises related to sources of self-efficacy beliefs: 1) mastery experiences, 2) vicarious experiences, 3) verbal persuasions, and 4) emotional and physiological states.

ELIGIBILITY:
Inclusion Criteria:

* Only psychiatric nurses.
* Still working at the time of data collection
* Willing to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2023-09-10 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Caring Efficacy | 3 months
  The Caring Efficacy Scale developed by Coates,3 is a 30-item, 6-point, Likert- type self-report scale (strongly disagree -3 to strongly agree +3), which assesses nurses' caring efficacy (i.e. confidence relating to ability to express a caring orientation and develop caring relationships with patients).
Psychiatric Nurses Job Stress | 3 months
  Psychiatric Nurses Job Stress Scale (PNJSS): was developed by Yada, (2011) and modified by Yada, (2015). It concerned with nurses' stressors in psychiatry departments by contributing to the self-care of psychiatric nurses and the line care of managerial staff. it containing 22 items.
perceived stigma | 3 months
  Perceived devaluation and discrimination scale (PDD): is a 12-item tool which measures the extent to which a person believes that most people will devalue or discriminate against someone with a mental illness. PDD was measured on a 4-point Likert scale with possible scores ranging from 1 to 4 agreement scale (1 = strongly disagree, 2 = disagree, 3 = agree, and 4 = strongly agree)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No